CLINICAL TRIAL: NCT02949037
Title: Enhancing mHealth Technology in the PCMH Environment to Activate Chronic Care Patients
Brief Title: Enhancing mHealth Technology to Activate Chronic Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clemson University (Other)
Collaborators: Madigan Army Medical Center (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB2015-234 (PPN 2015000085)
Record Dates: First submitted 2016-09-30; First posted 2016-10-31 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Use of (4) bluetooth-enabled biomedical devices (i.e. scale, blood pressure cuff, activity monitor, glucose monitor), for use in self care activities, integrated with the mobile health care environment (MHCE) system. The MHCE system will provide tailored behavioral messages triggered by clinical values and survey responses.
  Interventions: Other: Mobile Health Care Environment (MHCE)
- Control (No Intervention): Use of (4) bluetooth-enabled biomedical devices (i.e. scale, blood pressure cuff, activity monitor, glucose monitor), for use in self care activities, NOT integrated with the mobile health care environment (MHCE) system.

INTERVENTIONS:
Other: Mobile Health Care Environment (MHCE) — An integrated mobile health system modified to support type 2 diabetes self-care activities. Primary intervention includes visualization and trending of device outcomes AND tailored behavioral messages based on Patient Activation Measure scores.
  Other Names: mCare
  Arms: Intervention

SUMMARY:
Multi-site feasibility study designed to assist type-2 diabetes patients in self-care activities. The study includes Bluetooth-enabled medical devices (i.e. scales, blood pressure cuffs, glucometers, and activity monitors) for both intervention and control groups. Those in the intervention group will have the devices linked too a mobile health care environment that provides key benefits that include: device data trending, reinforcing tailored behavioral messages, and enhanced communication with the clinic.

DETAILED DESCRIPTION:
Multi-site phased study, conducted within the Military Health System that includes a user-centered design phase and a patient centered medical home (PCMH)-based feasibility trial.

In Phase I the investigators will assess both patient and clinician preferences and usability regarding the enhancement of the enabling technology capabilities for Type 2 diabetes chronic self-care management. The data from the experience will be coded and analyzed by the research team and the technology will be adapted accordingly before Phase II.

Phase II research is a single-blinded 12-month feasibility study that seeks to include the enabling technology to support diabetes self-care management with tailored behavioral messaging aimed at reinforcing and encouraging self-care behavior based on patients' readiness. We have included safety thresholds that alert patients and clinical team under certain conditions.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 years or older,
* Ability to understand and read English,
* Be empanelled to one of the target PCMH sites, and
* Diagnosed with type 2 diabetes.

Exclusion Criteria:

* pregnant women,
* non-English speaking patients,
* receiving hospice care,
* active cancer and treatment with chemotherapy or radiation therapy,
* taking Coumadin,
* recipient of gastric bypass or similar procedure,
* diagnosis of uncontrolled hypothyroidism,
* known Cushing's syndrome,
* being treated with oral steroids,
* known liver disease,
* current diagnosis of cognitive impairments which would interfere with use of technology,
* congestive heart failure New York Heart Association class 3 or 4,
* inability to use a mobile device due to cognitive or physical impairments, and
* PAM® score = 4 during initial screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure (PAM) | Every 3 months during the 12-month trial
  PAM is a validated survey measure of patient activation

SECONDARY OUTCOMES:
Glycosylated hemoglobin (HbA1C) | Every 4 months during 12-month trial
  HbA1c results documented on three occasions
Low-density Lipoprotein (LDL) | Every 4 months during 12-month trial
  LDL results documented on three occasions
High-density Lipoprotein (HDL) | Every 4 months during 12-month trial
  HDL results documented on three occasions
Abdominal circumference | Every 4 months during 12-month trial
  Abdominal measures taken on three occasions
Blood pressure | Every 4 months plus patient self-measurement during 12 -month trial
  Collected in clinic and daily by the patient
Summary of Diabetes Self-Care Activities (SDSCA) | Every 2 weeks during 12-month trial
  Validated survey measure of diabetes self-care activities

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W. Gimbel, Principal Investigator — Clemson University
Locations (2):
- United States (2):
  - Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada
  - Madigan Army Medicall Center, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gimbel RW, Rennert LM, Crawford P, Little JR, Truong K, Williams JE, Griffin SF, Shi L, Chen L, Zhang L, Moss JB, Marshall RC, Edwards KW, Crawford KJ, Hing M, Schmeltz A, Lumsden B, Ashby M, Haas E, Palazzo K. Enhancing Patient Activation and Self-Management Activities in Patients With Type 2 Diabetes Using the US Department of Defense Mobile Health Care Environment: Feasibility Study. J Med Internet Res. 2020 May 26;22(5):e17968. doi: 10.2196/17968. PMID 32329438
- [Derived] Gimbel R, Shi L, Williams JE, Dye CJ, Chen L, Crawford P, Shry EA, Griffin SF, Jones KO, Sherrill WW, Truong K, Little JR, Edwards KW, Hing M, Moss JB. Enhancing mHealth Technology in the Patient-Centered Medical Home Environment to Activate Patients With Type 2 Diabetes: A Multisite Feasibility Study Protocol. JMIR Res Protoc. 2017 Mar 6;6(3):e38. doi: 10.2196/resprot.6993. PMID 28264792

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT02949037/Prot_SAP_000.pdf